CLINICAL TRIAL: NCT02718027
Title: Biomarker for Alport Syndrome: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarker for Alport Syndrome (BioAlport)
Acronym: BioAlport
Status: Terminated | Type: Observational
Why Stopped: Study no longer pursued.
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BAP 06-2018
Record Dates: First submitted 2015-11-10; First posted 2016-03-24 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Nephritis, Hereditary; Hematuria-Nephropathy-Deafness Syndrome
Keywords: Alport Syndrome; Biomarker
MeSH Terms: conditions — Nephritis, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Alport Syndrome: Participants diagnosed with Alport syndrome aged between 2 months and 50 years

SUMMARY:
International, multicenter, observational, longitudinal monitoring study to identify biomarker/s for Alport syndrome and to explore the clinical robustness, specificity, and long-term variability of these biomarker/s

DETAILED DESCRIPTION:
Alport syndrome (AS) is a progressive hereditary glomerular disease with the prevalence 1 in 50,000. AS is caused by pathogenic variants in the COL4A3, COL4A4, and COL4A5 genes encoding type IV collagen α3, α4, and α5 chains, respectively. There are three modes of inheritance: X-linked Alport syndrome (XLAS), autosomal recessive AS (ARAS), and autosomal dominant AS (ADAS).

Alport Syndrome causes progressive kidney damage. The glomeruli and other normal kidney structures such as tubules are gradually replaced by scar tissue, leading to kidney failure. Boys with Alport Syndrome, regardless of the genetic type, eventually develop kidney failure. These boys often need dialysis or transplantation during their teenage or young adult years, but kidney failure can occur as late as 40-50 years of age in some men with Alport Syndrome. Most girls with the X-linked type of Alport Syndrome do not develop kidney failure. However, as women with Alport Syndrome get older the risk of kidney failure increases.

Currently, diagnosis of Alport Syndrome relies on careful evaluation of the patient's signs and symptoms, along with the family history. Hearing and vision should also be tested. The evaluation can also include a blood test, urine tests, and a kidney biopsy to determine Alport Syndrome. A genetic test is crucial to confirm the diagnosis and determine the genetic type of Alport Syndrome.

There is no cure for Alport syndrome; however, symptomatic treatment can help relieve symptoms. Kidney transplantation is usually very successful in people with Alport Syndrome and is considered the best treatment when end-stage kidney failure is approaching.

The aim of this study to identify biomarker/s for Alport Syndrome and to explore their clinical robustness, specificity, and long-term variability, in the attempt to offer access to earlier diagnosis and treatment monitoring.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent is obtained from the participant or the parent/ legal guardian.
* The participant is aged between 2 months and 50 years
* The diagnosis of Alport Syndrome is genetically confirmed by CENTOGENE

EXCLUSION CRITERIA

* Informed consent is not obtained from the participant or from the parent/ legal guardian
* The participant is younger than 2 months or older than 50 years
* The diagnosis of Alport Syndrome is not genetically confirmed by CENTOGENE

Ages: 2 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with Alport Syndrome
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of Alport Syndrome biomarker/s | 36 months
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and long-term variability of Alport syndrome biomarker/s | 36 months
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — Centogene GmbH
Locations (7):
- University Hospital Center Mother Teresa, Tirana, Albania
- Department of Molecular and Medical Genetics, Tbilisi State Medical University, Tbilisi, Georgia
- Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala, India
- Rare diseases coordinating centre, Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania
- Department of Pediatric Gastroenterology and Hepatology, The Children's Hospital and Institute of Child Health, Lahore, Pakistan
- Emergency Hospital for Children "Louis Turcanu", Timișoara, Romania
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided